CLINICAL TRIAL: NCT05056103
Title: Effect of an Automated Secretion Removal Technology, Named TrachFlush, on the Need for Tracheal Suctioning - Protocol for a Study in Intubated and Mechanically Ventilated Intensive Care Unit Patients
Brief Title: Automated Secretion Removal in ICU Patients
Acronym: TrachFlush
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Lack of financial support
Sponsor: Academisch Medisch Centrum - Universiteit van Amsterdam (AMC-UvA) (Other)
Responsible Party: Principal Investigator, Prof. Dr. Marcus J. Schultz, Prof., Academisch Medisch Centrum - Universiteit van Amsterdam (AMC-UvA)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: TrachFlush
Record Dates: First submitted 2021-09-15; First posted 2021-09-24 (Actual); Last update posted 2022-07-25 (Actual); Status verified 2022-07

CONDITIONS: Mechanical Ventilation Complication

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- TrachFlush (Other)
  Interventions: Device: TrachFlush

INTERVENTIONS:
Device: TrachFlush — The attending nurses activate the TrachFlush when there are secretions present in the larger airways that need to be removed. If this results into a push of airway secretions past and above the cuff of the endotracheal tube, no further action is needed. If unsuccessful, the nurse will perform a standard tracheal suctioning procedure to remove the secretions. In a subset of patients with an endotracheal tube that allows subglottal suctioning, the exact amount of airway secretions present above the cuff will be measured each time the TrachFlush is used.
  Other Names: endotracheal suctioning

SUMMARY:
SUMMARY Rationale In intubated and mechanically ventilated critically ill patients, removal of airway secretions is typically performed by tracheal suctioning, an intervention that is labor-intensive and very unpleasant for the patient. The current study tests the hypothesis that a novel secretion removal technology named TrachFlush, that pushes airway secretions past and above the cuff of the endotracheal tube, reduces the need for tracheal suctioning.

Objective The primary objective of this study is to evaluate whether use of the TrachFlush reduces the need for tracheal suctioning. In a selection of patients, one secondary objective is to ascertain the exact volume of airway secretions that is pushed past and above the cuff of the endotracheal tube.

Study design Open prospective intervention study. Study population One hundred adult, intubated and mechanically ventilated ICU patients expected to need invasive ventilation > 24 hours.

Intervention The attending nurses activate the TrachFlush when there are secretions present in the larger airways that need to be removed. If this results into a push of airway secretions past and above the cuff of the endotracheal tube, no further action is needed. If unsuccessful, the nurse will perform a standard tracheal suctioning procedure to remove the secretions. In a subset of patients with an endotracheal tube that allows subglottal suctioning, the exact amount of airway secretions present above the cuff will be measured each time the TrachFlush is used.

Main study parameters/endpoints The proportion of successful TrachFlush activations from start of the study to complete weaning from the ventilator, or a maximum of 7 days (primary). Secondary endpoints include the total number of TrachFlush activations during the same time window (all patients), and the exact amount of airway secretions pushed past and above the cuff of the endotracheal tube (in patients with a tube allows subglottal suctioning).

Nature and extent of the burden and risks associated with participation, benefit and group relatedness Inappropriate deflation or inflation of the endotracheal cuff by the TrachFlush could cause harm. However, the cuff pressure will be checked regularly, and if necessary corrected, at least every time the TrachFlush has been used. Patients may benefit from the intervention, as the need for tracheal suctioning may reduce.

ELIGIBILITY:
Inclusion Criteria:

* admission to one of the participating ICUs;
* intubated with an endotracheal tube containing a cuff;
* receiving invasive mechanical ventilation; and
* expected to need invasive ventilation beyond the following calendar day at the moment of inclusion.

Exclusion Criteria:

* age < 18 years;
* known or suspected tracheal damage, e.g., after inhalation trauma, thorax trauma, or intubation trauma;
* any condition for which deflation of the endotracheal cuff is deemed detrimental, e.g., in case high airway pressures are needed; and
* any infection, or colonization with pathogens that require strict single isolation of the patient (cohort isolation is allowed).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 28 (Actual)
Dates: Start 2021-09-15 (Actual); Primary Completion 2022-05-31 (Actual); Study Completion 2022-06-30 (Actual)

PRIMARY OUTCOMES:
proportion of successful TrachFlush activations from start of the study to complete weaning from the ventilator, or a maximum of 7 days | 7 days

SECONDARY OUTCOMES:
total number of TrachFlush activations during the same time window (all patients) | 7 days
incidence of hypoxemia related to the TrachFlush activation or tracheal suction | 7 days
Incidence of hypotension related to the TrachFlush activation or tracheal suction | 7 days
Incidence of patient agitation related to the TrachFlush activation or tracheal suctions | 7 days
The volume of subglottal secretions with each TrachFlush intervention (in a patients with an endotracheal tube in place that allows subglottic suctioning). | 7days

CONTACTS AND LOCATIONS:
Overall Officials: Frederique Paulus, PhD, Principal Investigator — AIDS Malignancy Consortium
Locations (1):
- Amsterdam UMC, Amsterdam, Netherlands

IPD SHARING:
Plan to Share IPD: Undecided